CLINICAL TRIAL: NCT02634983
Title: A Randomized, Double-blind, Placebo-controlled, Two-period Crossover Study to Assess the Effect of Inhaled QVA149 on Global and Regional Lung Function and Gas Exchange in Patients With Moderate to Severe COPD
Brief Title: QVA Mechanistic Efficacy Study (Receptor Effects, Etc)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2325; 2013-004461-13 (EudraCT Number)
Record Dates: First submitted 2015-10-28; First posted 2015-12-18 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Smokers; Ex-smokers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation | interventions — indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 110/50 mcg then Matching placebo (Experimental): Single daily dose of 110/50 μg QVA149 for 8-10 days.
  Interventions: Drug: QVA149
- Matching placebo then QVA149 110/50 mcg (Placebo Comparator): Single daily dose of matching placebo for 8-10 days.
  Interventions: Drug: QVA149; Drug: Placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 μg o.d. capsules for inhalation, supplied in blisters via the Concept 1 inhalation device, a single dose dry powder inhaler.
Drug: Placebo — Matching placebo
  Arms: Matching placebo then QVA149 110/50 mcg

SUMMARY:
The purpose of this study was to assess global ventilated lung volume in moderate to severe COPD patients using MRI lung imaging after treatment with QVA149 compared to placebo.

DETAILED DESCRIPTION:
The MRI approach represented an opportunity to better understand the impact of a potent dual bronchodilator on the small and central airways and thereby increasing ventilated lung volume, gas exchange, and ventilation-perfusion deficits.

The study investigated the effect of QVA149 on global and regional lung ventilation using MRI lung imaging to enhance the understanding of QVA pharmacology in COPD patients.

ELIGIBILITY:
Key Inclusion Criteria:

Males and females with COPD aged 40 years and above, weighing ≥45 kg and ≤100 kg, who were smokers and ex-smokers who had a smoking history of at least 10 pack years, and diagnosed with moderate to severe COPD according to GOLD 2015 criteria were included in the study. Patients with airflow limitation indicated by a post-bronchodilator FEV1/FVC < 0.70 and by a post-bronchodilator FEV1 ≥ 30 % and <80 % were included in the study. Post-bronchodilator refers to 1 hr (+/- 5 minutes) after sequential inhalation of 84 µg ipratropium bromide (or equivalent dose) and 400 µg salbutamol/360 µg albuterol (or equivalent dose).

Key Exclusion Criteria:

Patients with conditions which could compromise patient safety and compliance (as judged by the investigator), as well as conditions that required oxygen therapy for chronic hypoxemia, ≥25% emphysematous changes on a scan within 6 months to screening, those with lower respiratory infections within 6 weeks of screening, and patients with concomitant pulmonary disease were excluded from the study. Patients with asthma were also excluded from the study.

Pregnant or nursing (lactating) women, patients with poorly controlled Type I or Type II diabetes, patients with poor renal function, and those who were unable to use a dry powder inhaler or perform spirometry, and had contraindications to MRI were also excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United Kingdom (3):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh D, Wild JM, Saralaya D, Lawson R, Marshall H, Goldin J, Brown MS, Kostikas K, Belmore K, Fogel R, Patalano F, Drollmann A, Machineni S, Jones I, Yates D, Tillmann HC. Effect of indacaterol/glycopyrronium on ventilation and perfusion in COPD: a randomized trial. Respir Res. 2022 Feb 10;23(1):26. doi: 10.1186/s12931-022-01949-3. PMID 35144620
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in 3 clinical sites in United-Kingdom
Pre-assignment Details: 31 patients were randomized, all of whom were included in the safety set and PD analysis sets (primary population of interest)
Groups:
- QVA149 110/50 mcg Then Matching Placebo: QVA149, followed by matching placebo. Each treatment 8-10 days.
- Matching Placebo Then QVA149 110/50 mcg: Matching placebo, followed by QVA149. Each treatment 8-10 days.
Period: Period One (First Treatment, 8-10 Days)
Arm/Group | QVA149 110/50 mcg Then Matching Placebo | Matching Placebo Then QVA149 110/50 mcg
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Washout (Approximately 7-14 Days)
Arm/Group | QVA149 110/50 mcg Then Matching Placebo | Matching Placebo Then QVA149 110/50 mcg
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Period 2 (Second Treatment, 8-10 Days)
Arm/Group | QVA149 110/50 mcg Then Matching Placebo | Matching Placebo Then QVA149 110/50 mcg
Started | 16 | 15
Completed | 14 | 15
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either QVA149 110/50 mcg or Placebo matching QVA149 110/50 mcg
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Forced Expiratory Volume in 1 Second [Mean (Standard Deviation); unit: Liter] — Spirometry assessments are to be performed 60 minutes post short-acting β2-adrenergic agonist (SABA) and short-acting muscarinic antagonist (SAMA) inhalation as part of the Baseline assessments. The Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  Liter
    0 Minutes Pre Inhalation | 1.1584 (0.35206)
    60 Minutes Post Inhalation | 1.3987 (0.37266)
Percent Predicted FEV1 [Mean (Standard Deviation); unit: Percent] — Spirometry assessments are to be performed 60 minutes post short-acting β2-adrenergic agonist (SABA) and short-acting muscarinic antagonist (SAMA) inhalation as part of the Baseline assessments.
  Percent
    0 Minutes Pre Inhalation | 43.90 (10.873)
    60 Minutes Post Inhalation | 53.10 (11.680)
Forced Vital Capacity [Mean (Standard Deviation); unit: Liter] — Spirometry assessments are to be performed 60 minutes post short-acting β2-adrenergic agonist (SABA) and short-acting muscarinic antagonist (SAMA) inhalation as part of the Baseline assessments. Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry.
  Liter
    0 Minutes Pre Inhalation | 2.7426 (0.73932)
    60 Minutes Post Inhalation | 3.0781 (0.81113)
FEV1/FVC ratio [Mean (Standard Deviation); unit: Percent ((FEV1/FVC)*100)] — Spirometry assessments are to be performed 60 minutes post short-acting β2-adrenergic agonist (SABA) and short-acting muscarinic antagonist (SAMA) inhalation as part of the Baseline assessments. The FEV1/FVC ratio is the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
  Percent ((FEV1/FVC)*100)
    0 Minutes Pre Inhalation | 42.968 (8.9797)
    60 Minutes Post Inhalation | 46.365 (8.8240)
Reversibility [Mean (Standard Deviation); unit: Liter] — Reversibility = FEV1 post-inhalation - FEV1 pre-inhalation. Reversibility was reported in absolute FEV1 values pre- and post-bronchodilator.
  Liter | 0.2403 (0.12994)
Reversibility [Mean (Standard Deviation); unit: Percent] — Reversibility = FEV1 post-inhalation - FEV1 pre-inhalation. Reversibility was reported in change in FEV1 between pre- and postbronchodilator assessment expressed in % of pre-bronchodilator FEV1.
  Percent | 9.19 (4.743)

OUTCOME MEASURES:

1. Primary Outcome: Global Ventilated Lung Volume
Description: The global distribution of inhaled gas within the lung was assessed using an inhaled gaseous contrast agent, Hyperpolarized Helium (3He) Lung Imaging. The Global Ventilated Lung Volume was expressed in percentage (%VV) of total lung volume.
Time Frame: Day 8 to Day 10 (each treatment period)
Population: The PD Analysis Set, which consisted of all participants with valid results assessed in each treatment period, was considered.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of total lung volume
Groups:
- QVA149 110/50 mcg: Single daily dose of 110/50 μg QVA149 for 8-10 days.
- Matching Placebo: Single daily dose of matching placebo for 8-10 days.
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 31 | 28
Percentage of total lung volume | 61.73 [56.16 to 67.30] | 56.73 [51.07 to 62.39]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; Global Ventilated Lung Volume; Test type: Non-Inferiority — Parameters were analyzed using mixed effects model including sequence, period, treatment as fixed factors and patient as random factor; p = 0.0254, t-test, 2 sided; Mean Difference (Final Values) = 5.00, 90% CI 2-sided [1.40 to 8.60], Standard Error of Mean 2.11

2. Secondary Outcome: Regional Ventilated Lung Volume
Description: The regional distribution of inhaled gas within the lung was assessed using an inhaled gaseous contrast agent, Hyperpolarized Helium (3He) Lung Imaging. The Regional Ventilated Lung Volume was expressed in percentage (% VDV) of total lung volume for each lobar region.
Time Frame: Day 8 to Day 10 (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of total lung volume
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 31 | 28
Percentage of total lung volume
  Lung, Left Ventilation | 61.94 [56.04 to 67.83] | 57.16 [51.17 to 63.15]
  Lung, Left Lower Lobe Ventilation | 58.97 [52.63 to 65.31] | 54.01 [47.52 to 60.49]
  Lung, Left Upper Lobe Ventilation | 64.17 [57.95 to 70.39] | 59.20 [52.87 to 65.53]
  Lung, Right Ventilation | 61.63 [55.90 to 67.36] | 56.24 [50.40 to 62.08]
  Lung, Right Lower Lobe Ventilation | 60.92 [54.62 to 67.21] | 57.65 [51.26 to 64.04]
  Lung, Right Middle Lobe Ventilation | 59.59 [52.85 to 66.34] | 53.98 [47.01 to 60.95]
  Lung, Right Upper Lobe Ventilation | 63.25 [56.71 to 69.79] | 55.53 [48.85 to 62.20]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0350, t-test, 2 sided; Mean Difference (Final Values) = 4.77, 90% CI 2-sided [1.11 to 8.44], Standard Error of Mean 2.15
Statistical Analysis 2: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Lower Lobe Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0946, t-test, 2 sided; Mean Difference (Final Values) = 4.96, 90% CI 2-sided [0.08 to 9.84], Standard Error of Mean 2.86
Statistical Analysis 3: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Upper Lobe Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0486, t-test, 2 sided; Mean Difference (Final Values) = 4.97, 90% CI 2-sided [0.87 to 9.07], Standard Error of Mean 2.41
Statistical Analysis 4: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0286, t-test, 2 sided; Mean Difference (Final Values) = 5.39, 90% CI 2-sided [1.42 to 9.35], Standard Error of Mean 2.33
Statistical Analysis 5: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Lower Lobe Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1650, t-test, 2 sided; Mean Difference (Final Values) = 3.27, 90% CI 2-sided [-0.63 to 7.17], Standard Error of Mean 2.29
Statistical Analysis 6: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Middle Lobe Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1421, t-test, 2 sided; Mean Difference (Final Values) = 5.61, 90% CI 2-sided [-0.71 to 11.94], Standard Error of Mean 3.71
Statistical Analysis 7: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Upper Lobe Ventilation; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0099, t-test, 2 sided; Mean Difference (Final Values) = 7.73, 90% CI 2-sided [2.98 to 12.47], Standard Error of Mean 2.78

3. Secondary Outcome: Pulmonary Perfusion
Description: Lung Perfusion Imaging, or MR perfusion imaging of the lung with gadolinium contrast agent, was performed to determine whether vascular abnormalities producing perfusion deficits corresponded to abnormalities in ventilation (hypoxic vasoconstriction). Pulmonary Perfusion was expressed in ml/100 g lung tissue/min of each lobar region.
Time Frame: Day 8 to Day 10 (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ml/100 g lung tissue/min
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 27 | 26
ml/100 g lung tissue/min
  Lung Perfusion | 13.96 [12.50 to 15.41] | 13.03 [11.56 to 14.50]
  Lung, Left Perfusion | 14.42 [12.94 to 15.90] | 13.08 [11.58 to 14.57]
  Lung, Left Lower Lobe Perfusion | 13.48 [11.91 to 15.06] | 12.79 [11.20 to 14.38]
  Lung, Left Upper Lobe Perfusion | 15.35 [13.69 to 17.01] | 13.45 [11.77 to 15.12]
  Lung, Right Perfusion | 13.54 [12.07 to 15.01] | 12.97 [11.49 to 14.46]
  Lung, Right Lower Lobe Perfusion | 13.26 [11.74 to 14.79] | 13.25 [11.71 to 14.79]
  Lung, Right Middle Lobe Perfusion | 14.86 [12.72 to 17.00] | 13.36 [11.19 to 15.53]
  Lung, Right Upper Lobe Perfusion | 13.57 [11.91 to 15.23] | 12.70 [11.03 to 14.37]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3230, t-test, 2 sided; Mean Difference (Final Values) = 0.93, 90% CI 2-sided [-0.64 to 2.50], Standard Error of Mean 0.92
Statistical Analysis 2: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1717, t-test, 2 sided; Mean Difference (Final Values) = 1.34, 90% CI 2-sided [-0.29 to 2.97], Standard Error of Mean 0.95
Statistical Analysis 3: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Lower Lobe Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5031, t-test, 2 sided; Mean Difference (Final Values) = 0.69, 90% CI 2-sided [-1.05 to 2.43], Standard Error of Mean 1.02
Statistical Analysis 4: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Left Upper Lobe Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0760, t-test, 2 sided; Mean Difference (Final Values) = 1.90, 90% CI 2-sided [0.15 to 3.65], Standard Error of Mean 1.03
Statistical Analysis 5: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5465, t-test, 2 sided; Mean Difference (Final Values) = 0.57, 90% CI 2-sided [-1.02 to 2.16], Standard Error of Mean 0.93
Statistical Analysis 6: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Lower Lobe Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.9913, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-1.85 to 1.87], Standard Error of Mean 1.08
Statistical Analysis 7: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Middle Lobe Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3837, t-test, 2 sided; Mean Difference (Final Values) = 1.51, 90% CI 2-sided [-1.39 to 4.40], Standard Error of Mean 1.70
Statistical Analysis 8: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung, Right Upper Lobe Perfusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3624, t-test, 2 sided; Mean Difference (Final Values) = 0.87, 90% CI 2-sided [-0.73 to 2.48], Standard Error of Mean 0.94

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: The Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
Time Frame: Day 1 (0.25, 1 and 2 hours post-dose), Day 8 (-0.75, -0.25, 0.25, 1 and 2 hours post-dose) (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liter
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 31 | 31
Liter
  FEV1 Day 1 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 29
  FEV1 Day 1 (0.25 hrs post-dose) | 1.27 [1.25 to 1.30] | 1.13 [1.10 to 1.15]
  FEV1 Day 1 (1 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1 Day 1 (1 hrs post-dose) | 1.32 [1.29 to 1.36] | 1.12 [1.09 to 1.16]
  FEV1 Day 1 (2 hrs post-dose): number analyzed (Participants) | 31 | 30
  FEV1 Day 1 (2 hrs post-dose) | 1.34 [1.30 to 1.38] | 1.15 [1.11 to 1.19]
  FEV1 Day 8 (-0.75 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1 Day 8 (-0.75 hrs post-dose) | 1.30 [1.26 to 1.34] | 1.09 [1.05 to 1.13]
  FEV1 Day 8 (-0.25 hrs post-dose): number analyzed (Participants) | 30 | 27
  FEV1 Day 8 (-0.25 hrs post-dose) | 1.33 [1.29 to 1.37] | 1.11 [1.07 to 1.15]
  FEV1 Day 8 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1 Day 8 (0.25 hrs post-dose) | 1.38 [1.35 to 1.42] | 1.10 [1.06 to 1.14]
  FEV1 Day 8 (1 hrs post-dose): number analyzed (Participants) | 30 | 26
  FEV1 Day 8 (1 hrs post-dose) | 1.45 [1.41 to 1.49] | 1.13 [1.09 to 1.17]
  FEV1 Day 8 (2 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1 Day 8 (2 hrs post-dose) | 1.43 [1.39 to 1.47] | 1.11 [1.07 to 1.15]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 1 (0.25 hrs post-dose); Test type: Non-Inferiority — Parameters were analyzed using mixed effects model including sequence, period, treatment, time and treatment*Day*time interaction term as fixed factors and patient factor as random factor. Day*time was repeated within each patient*period interaction and subject average baseline and period adjusted baseline were included as covariates; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [0.11 to 0.18], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 1 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.20, 90% CI 2-sided [0.15 to 0.25], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 1 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [0.13 to 0.24], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 8 (-0.75 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.22, 90% CI 2-sided [0.16 to 0.27], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 8 (-0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.22, 90% CI 2-sided [0.16 to 0.28], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 8 (0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [0.23 to 0.33], Standard Error of Mean 0.03
Statistical Analysis 7: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 8 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.32, 90% CI 2-sided [0.26 to 0.37], Standard Error of Mean 0.03
Statistical Analysis 8: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1 Day 8 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.32, 90% CI 2-sided [0.26 to 0.38], Standard Error of Mean 0.04

5. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. An increase in FVC indicates improvement in lung function.
Time Frame: Day 1 (0.25, 1 and 2 hours post-dose), Day 8 (-0.75, -0.25, 0.25, 1 and 2 hours post-dose) (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liter
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 31 | 31
Liter
  FVC Day 1 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 29
  FVC Day 1 (0.25 hrs post-dose) | 2.92 [2.85 to 2.98] | 2.68 [2.61 to 2.74]
  FVC Day 1 (1 hrs post-dose): number analyzed (Participants) | 31 | 28
  FVC Day 1 (1 hrs post-dose) | 2.99 [2.91 to 3.06] | 2.63 [2.56 to 2.71]
  FVC Day 1 (2 hrs post-dose): number analyzed (Participants) | 31 | 30
  FVC Day 1 (2 hrs post-dose) | 2.99 [2.91 to 3.07] | 2.68 [2.59 to 2.76]
  FVC Day 8 (-0.75 hrs post-dose): number analyzed (Participants) | 31 | 28
  FVC Day 8 (-0.75 hrs post-dose) | 2.91 [2.84 to 2.98] | 2.56 [2.49 to 2.64]
  FVC Day 8 (-0.25 hrs post-dose): number analyzed (Participants) | 30 | 27
  FVC Day 8 (-0.25 hrs post-dose) | 2.91 [2.84 to 2.98] | 2.63 [2.56 to 2.70]
  FVC Day 8 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 28
  FVC Day 8 (0.25 hrs post-dose) | 3.02 [2.95 to 3.09] | 2.59 [2.51 to 2.66]
  FVC Day 8 (1 hrs post-dose): number analyzed (Participants) | 30 | 26
  FVC Day 8 (1 hrs post-dose) | 3.10 [3.04 to 3.17] | 2.65 [2.58 to 2.72]
  FVC Day 8 (2 hrs post-dose): number analyzed (Participants) | 31 | 28
  FVC Day 8 (2 hrs post-dose) | 3.06 [2.98 to 3.13] | 2.62 [2.54 to 2.70]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 1 (0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.24, 90% CI 2-sided [0.15 to 0.33], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 1 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.35, 90% CI 2-sided [0.25 to 0.45], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 1 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.31, 90% CI 2-sided [0.20 to 0.42], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 8 (-0.75 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 0.35, 90% CI 2-sided [0.25 to 0.45], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 8 (-0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [0.19 to 0.37], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 8 (0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.43, 90% CI 2-sided [0.33 to 0.53], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 8 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [0.36 to 0.54], Standard Error of Mean 0.06
Statistical Analysis 8: Comparison: QVA149 110/50 mcg vs Matching Placebo; FVC Day 8 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.44, 90% CI 2-sided [0.33 to 0.55], Standard Error of Mean 0.06

6. Secondary Outcome: FEV1/FVC Ratio
Description: The FEV1/FVC ratio is the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC). The result of this ratio is expressed as FEV1%.
Time Frame: Day 1 (0.25, 1 and 2 hours post-dose), Day 8 (-0.75, -0.25, 0.25, 1 and 2 hours post-dose) (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: FEV1 Percentage
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 31 | 31
FEV1 Percentage
  FEV1/FVC Day 1 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 29
  FEV1/FVC Day 1 (0.25 hrs post-dose) | 44.31 [43.59 to 45.02] | 42.14 [41.39 to 42.89]
  FEV1/FVC Day 1 (1 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1/FVC Day 1 (1 hrs post-dose) | 44.97 [44.05 to 45.88] | 42.91 [41.95 to 43.87]
  FEV1/FVC Day 1 (2 hrs post-dose): number analyzed (Participants) | 31 | 30
  FEV1/FVC Day 1 (2 hrs post-dose) | 45.25 [44.42 to 46.08] | 42.93 [42.08 to 43.79]
  FEV1/FVC Day 8 (-0.75 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1/FVC Day 8 (-0.75 hrs post-dose) | 45.05 [44.05 to 46.05] | 42.23 [41.16 to 43.30]
  FEV1/FVC Day 8 (-0.25 hrs post-dose): number analyzed (Participants) | 30 | 27
  FEV1/FVC Day 8 (-0.25 hrs post-dose) | 45.97 [45.05 to 46.89] | 42.17 [41.19 to 43.15]
  FEV1/FVC Day 8 (0.25 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1/FVC Day 8 (0.25 hrs post-dose) | 46.34 [45.43 to 47.26] | 42.60 [41.63 to 43.58]
  FEV1/FVC Day 8 (1 hrs post-dose): number analyzed (Participants) | 30 | 26
  FEV1/FVC Day 8 (1 hrs post-dose) | 47.32 [46.31 to 48.33] | 42.72 [41.64 to 43.80]
  FEV1/FVC Day 8 (2 hrs post-dose): number analyzed (Participants) | 31 | 28
  FEV1/FVC Day 8 (2 hrs post-dose) | 47.39 [46.39 to 48.40] | 42.42 [41.35 to 43.48]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 1 (0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.0006, t-test, 2 sided; Mean Difference (Final Values) = 2.17, 90% CI 2-sided [1.21 to 3.12], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 1 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.0106, t-test, 2 sided; Mean Difference (Final Values) = 2.06, 90% CI 2-sided [0.78 to 3.33], Standard Error of Mean 0.75
Statistical Analysis 3: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 1 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.0013, t-test, 2 sided; Mean Difference (Final Values) = 2.32, 90% CI 2-sided [1.20 to 3.44], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 8 (-0.75 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.0017, t-test, 2 sided; Mean Difference (Final Values) = 2.82, 90% CI 2-sided [1.41 to 4.23], Standard Error of Mean 0.83
Statistical Analysis 5: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 8 (-0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.80, 90% CI 2-sided [2.51 to 5.09], Standard Error of Mean 0.76
Statistical Analysis 6: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 8 (0.25 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.74, 90% CI 2-sided [2.45 to 5.02], Standard Error of Mean 0.75
Statistical Analysis 7: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 8 (1 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 4.60, 90% CI 2-sided [3.16 to 6.03], Standard Error of Mean 0.85
Statistical Analysis 8: Comparison: QVA149 110/50 mcg vs Matching Placebo; FEV1/FVC Day 8 (2 hrs post-dose); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 4.98, 90% CI 2-sided [3.56 to 6.39], Standard Error of Mean 0.83

7. Secondary Outcome: Lung Clearance Index by Multiple Breath Nitrogen Washout (MBNW)
Description: Multiple Breath Nitrogen Washout (MBNW) was performed after 2 hours post-dose spirometry assessments using a multiple breath inert gas washout technique. The device provides the global index of ventilation inhomogeneity assessment (LCI = Cumulative Expired Volume/Functional Residual Capacity).
Time Frame: Day 8 (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 29 | 26
Ratio | 10.80 [10.22 to 11.37] | 10.81 [10.20 to 11.41]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; Lung Clearance Index; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.9820, t-test, 2 sided; Mean Difference (Final Values) = -0.01, 90% CI 2-sided [-0.62 to 0.60], Standard Error of Mean 0.36

8. Secondary Outcome: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: The diffusing capacity of the lung for carbon monoxide (DLCO) is a measure of how easily carbon monoxide (CO) molecules transfer from the alveolar gas to the hemoglobin of the red cells in the pulmonary circulation. To measure the DLCO, the patient inhales a single breath containing a minute amount of CO and holds it for 10 seconds. The breath is then exhaled and the exhaled breath is analyzed for CO. The change in the concentration of the CO is then multiplied by the single breath TLC to calculate the DLCO.
Time Frame: Day 8 (each treatment period)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mL/min/mmHg
Arm/Group | QVA149 110/50 mcg | Matching Placebo
Number analyzed (Participants) | 29 | 26
mL/min/mmHg | 16.38 [14.77 to 18.00] | 15.73 [14.10 to 17.35]
Statistical Analysis 1: Comparison: QVA149 110/50 mcg vs Matching Placebo; Diffusion Capacity of Lung for CO; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0821, t-test, 2 sided; Mean Difference (Final Values) = 0.66, 90% CI 2-sided [0.04 to 1.27], Standard Error of Mean 0.36

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 1 year.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Arm/Group | QVA149 110/50 mcg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/31
Other Adverse Events (participants affected / at risk) | 5/31 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110/50 mcg (N=31) | Matching Placebo (N=31)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110/50 mcg (N=31) | Matching Placebo (N=31)
Vomiting (Gastrointestinal disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02634983/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02634983/SAP_001.pdf